CLINICAL TRIAL: NCT00082433
Title: A Phase III Study of Novel Epothilone (Ixabepilone) Plus Capecitabine Versus Capecitabine Alone in Patients With Advanced Breast Cancer Previously Treated With an Anthracycline and a Taxane
Brief Title: Epothilone (Ixabepilone) Plus Capecitabine Versus Capecitabine Alone in Patients With Advanced Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: R-Pharm (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA163-048
Record Dates: First submitted 2004-05-07; First posted 2004-05-11 (Estimated); Results first posted 2009-08-17 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Cancer; Breast Cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms | interventions — ixabepilone; Capecitabine; Epothilones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Ixabepilone + Capecitabine
- B (Active Comparator)
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Ixabepilone + Capecitabine — Ixabepilone lypholized powder/Diluent for solution for injection/Tablets, IV/Oral, 40 mg/m2 + Capecitabine 2000 mg/m2, Ixabepilone on Day 1 and Capecitabine twice daily Days 1-14 of 21 day cycle
  Other Names: IXEMPRA®; Epothilone
  Arms: A
Drug: Capecitabine — Tablet, Oral, 2500 mg/m2, Capecitabine twice daily Days 1-14 of 21 day cycle
  Arms: B

SUMMARY:
The purpose of this clinical research study is to learn if BMS-247550 added to the approved therapy of capecitabine (Xeloda) provides measurable clinical benefits over capecitabine alone in women with metastatic breast cancer. Patients should have previously received an anthracycline and a taxane. The safety of this treatment will also be studied.

ELIGIBILITY:
* Patients must have received prior treatment which included both an anthracycline (i.e., doxorubicin or epirubicin) and a taxane (i.e., paclitaxel or docetaxel).
* Patients must have received no more than two prior chemotherapy regimens. Patients who have not received treatment for metastatic disease must have relapsed within one year.
* Patients may not have any history of brain and/or leptomeningeal metastases.
* Patients may not have Grade 2 or worse neuropathy at the time of study entry.
* Patients may not have had prior treatment with any epothilones and/or capecitabine (i.e. Xeloda)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1221 (Actual)
Dates: Start 2003-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (186):
- United States (34):
  - Local Institution, Tucson, Arizona
  - Local Institution, Beverly Hills, California
  - Local Institution, Corona, California
  - Local Institution, Hartford, Connecticut
  - Local Institution, Plantation, Florida
  - Local Institution, Boise, Idaho
  - Local Institution, Evanston, Illinois
  - Local Institution, Iowa City, Iowa
  - Local Institution, Louisville, Kentucky
  - Local Institution, Baton Rouge, Louisiana
  - Local Institution, Bethesda, Maryland
  - Local Institution, Boston, Massachusetts
  - Local Institution, Jackson, Mississippi
  - Local Institution, Columbia, Missouri
  - Local Institution, Voorhees Township, New Jersey
  - Local Institution, Albuquerque, New Mexico
  - Local Institution, Latham, New York
  - Local Institution, Mineola, New York
  - Local Institution, New York, New York
  - Local Institution, The Bronx, New York
  - Local Institution, Durham, North Carolina
  - Local Institution, Goldsboro, North Carolina
  - Local Institution, Hickory, North Carolina
  - Local Institution, Kinston, North Carolina
  - Local Institution, Canton, Ohio
  - Local Institution, Columbus, Ohio
  - Local Institution, Langhorne, Pennsylvania
  - Local Institution, Knoxville, Tennessee
  - Local Institution, Memphis, Tennessee
  - Local Institution, Dallas, Texas
  - Local Institution, Charlottesville, Virginia
  - Local Institution, Norfolk, Virginia
  - Local Institution, Richmond, Virginia
  - Local Institution, Marshfield, Wisconsin
- Argentina (11):
  - Local Institution, Avellaneda, Buenos Aires
  - Local Institution, Bahía Blanca, Buenos Aires
  - Local Institution, Belén de Escobar, Buenos Aires
  - Local Institution, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Local Institution, Resistencia, Chaco Province
  - Local Institution, Barrio Alto Verde, Córdoba Province
  - Local Institution, San Miguel de Tucumán, Tucumán Province
  - Local Institution, Buenos Aires
  - Local Institution, Mendoza
  - Local Institution, Salta
  - Local Institution, Santa Fe
- Australia (11):
  - Local Institution, Sydney, New South Wales
  - Local Institution, Westmead, New South Wales
  - Local Institution, Brisbane, Queensland
  - Local Institution, Herston, Queensland
  - Local Institution, South Brisbane, Queensland
  - Local Institution, Toowoomba, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Woodville, South Australia
  - Local Institution, East Melbourne, Victoria
  - Local Institution, Parkville, Victoria
  - Local Institution, Perth, Western Australia
- Austria (3):
  - Local Institution, Graz
  - Local Institution, Vienna
  - Local Institution, Vöcklabruck
- Belgium (6):
  - Local Institution, Brussels
  - Local Institution, Charleroi
  - Local Institution, Ghent
  - Local Institution, Hasselt
  - Local Institution, Kortrijk
  - Local Institution, Wilrijk
- Brazil (5):
  - Local Institution, Centro-Porto Alegre, Rio Grande do Sul
  - Local Institution, Bela Vista, São Paulo
  - Local Institution, Higienopolis, São Paulo
  - Local Institution, São Paulo, São Paulo
  - Local Institution, Rio de Janeiro
- Canada (2):
  - Local Institution, Thunder Bay, Ontario
  - Local Institution, Montreal, Quebec
- Local Institution, Santiago, Santiago Metropolitan, Chile
- China (9):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Nanjing, Jiangsu
  - Local Institution, Dalian, Liaoning
  - Local Institution, Dilian, Liaoning
  - Local Institution, Jinan, Shandong
  - Local Institution, Shanghai, Shanghai Municipality
  - Local Institution, Xi’an, Shanxi
  - Local Institution, Hangzhou, Zhejiang
- Croatia (2):
  - Local Institution, Split
  - Local Institution, Zagreb
- Czechia (3):
  - Local Institution, Brno
  - Local Institution, Hradec Králové
  - Local Institution, Prague
- Denmark (3):
  - Local Institution, Aalborg
  - Local Institution, Herlev
  - Local Institution, København Ø
- France (15):
  - Local Institution, Angers
  - Local Institution, Bordeaux
  - Local Institution, Caen
  - Local Institution, Clermont-Ferrand
  - Local Institution, Colmar
  - Local Institution, Le Mans
  - Local Institution, Metz
  - Local Institution, Paris
  - Local Institution, Pierre-Bénite
  - Local Institution, Reims
  - Local Institution, Saint-Brieuc
  - Local Institution, Saint-Grégoire
  - Local Institution, Saint-Herblain
  - Local Institution, Tours
  - Local Institution, Villejuif
- Germany (13):
  - Local Institution, Berlin
  - Local Institution, Erlangen
  - Local Institution, Essen
  - Local Institution, Hanover
  - Local Institution, Karlsruhe
  - Local Institution, Kiel
  - Local Institution, Marburg
  - Local Institution, München
  - Local Institution, Rehling
  - Local Institution, Saarbrücken
  - Local Institution, Tübingen
  - Local Institution, Ulm
  - Local Institution, Wiesbaden
- Greece (4):
  - Local Institution, Athens
  - Local Institution, Crete
  - Local Institution, Pátrai
  - Local Institution, Thessaloniki
- Ireland (4):
  - Local Institution, Wilton, Cork
  - Local Institution, Cork
  - Local Institution, Dublin
  - Local Institution, Galway
- Israel (4):
  - Local Institution, Haifa
  - Local Institution, Jerusalem
  - Local Institution, Ramat Gan
  - Local Institution, Tel Aviv
- Italy (12):
  - Local Institution, Rozzano, Milan
  - Local Institution, Bari
  - Local Institution, Florence
  - Local Institution, Genova
  - Local Institution, Milan
  - Local Institution, Modena
  - Local Institution, Perugia
  - Local Institution, Potenza
  - Local Institution, Roma
  - Local Institution, San Giovanni Rotondo
  - Local Institution, Sora
  - Local Institution, Torino
- Netherlands (4):
  - Local Institution, Arnhem
  - Local Institution, Enschede
  - Local Institution, The Hague
  - Local Institution, Zwolle
- Portugal (2):
  - Local Institution, Coimbra
  - Local Institution, Lisbon
- Russia (3):
  - Local Institution, Kazan'
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- Local Institution, Singapore, Singapore
- South Africa (4):
  - Local Institution, Port Elizabeth, Eastern Cape
  - Local Institution, Johannesburg, Gauteng
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Panorama, Western Cape
- South Korea (3):
  - Local Institution, Gyeonggi-do
  - Local Institution, Incheon
  - Local Institution, Seoul
- Spain (15):
  - Local Institution, Terassa, Barcelona
  - Local Institution, Barcelona
  - Local Institution, Cadiz
  - Local Institution, Córdoba
  - Local Institution, Elche (Alicante)
  - Local Institution, Jaén
  - Local Institution, L'Hospitalet de Llobregat
  - Local Institution, Madrid
  - Local Institution, Pontevedra
  - Local Institution, Reus
  - Local Institution, Salamanca
  - Local Institution, Santa Cruz de Tenerife
  - Local Institution, Seville
  - Local Institution, Valencia
  - Local Institution, Zaragoza
- Switzerland (3):
  - Local Institution, Bern
  - Local Institution, Thun
  - Local Institution, Zurich
- Local Institution, Taipei, Taiwan
- Turkey (Türkiye) (3):
  - Local Institution, Ankara
  - Local Institution, Istanbul
  - Local Institution, Izmir
- United Kingdom (5):
  - Local Institution, Belfast, Armagh
  - Local Institution, Glasgow, Central
  - Local Institution, London, Greater London
  - Local Institution, Shrewsbury, Shropshire
  - Local Institution, Birmingham, West Midlands

REFERENCES:
- [Derived] Wedam SB, Beaver JA, Amiri-Kordestani L, Bloomquist E, Tang S, Goldberg KB, Sridhara R, Ibrahim A, Kim G, Kluetz P, McKee A, Pazdur R. US Food and Drug Administration Pooled Analysis to Assess the Impact of Bone-Only Metastatic Breast Cancer on Clinical Trial Outcomes and Radiographic Assessments. J Clin Oncol. 2018 Apr 20;36(12):1225-1231. doi: 10.1200/JCO.2017.74.6917. Epub 2018 Mar 9. PMID 29522361
- [Derived] Vahdat LT, Vrdoljak E, Gomez H, Li RK, Bosserman L, Sparano JA, Baselga J, Mukhopadhyay P, Valero V. Efficacy and safety of ixabepilone plus capecitabine in elderly patients with anthracycline- and taxane-pretreated metastatic breast cancer. J Geriatr Oncol. 2013 Oct;4(4):346-52. doi: 10.1016/j.jgo.2013.07.006. Epub 2013 Aug 23. PMID 24472478
- [Derived] Jassem J, Fein L, Karwal M, Campone M, Peck R, Poulart V, Vahdat L. Ixabepilone plus capecitabine in advanced breast cancer patients with early relapse after adjuvant anthracyclines and taxanes: a pooled subset analysis of two phase III studies. Breast. 2012 Feb;21(1):89-94. doi: 10.1016/j.breast.2011.09.003. Epub 2011 Sep 21. PMID 21937232
- [Derived] Roche H, Conte P, Perez EA, Sparano JA, Xu B, Jassem J, Peck R, Kelleher T, Hortobagyi GN. Ixabepilone plus capecitabine in metastatic breast cancer patients with reduced performance status previously treated with anthracyclines and taxanes: a pooled analysis by performance status of efficacy and safety data from 2 phase III studies. Breast Cancer Res Treat. 2011 Feb;125(3):755-65. doi: 10.1007/s10549-010-1251-y. Epub 2010 Dec 3. PMID 21128114

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: PLEASE NOTE: Completed=number of participants completing ≥18 cycles of treatment; not completed=number of subjects coming off study treatment prior to completing at least 18 cycles, with specified reasons for coming off study treatment. Participants continued to be followed for overall survival.
Groups:
- Ixabepilone + Capecitabine: Ixabepilone in combination with capecitabine (combination group): Ixabepilone 40 mg/m2 administered as a 3-hour intravenous (IV) infusion on Day 1 of each cycle only, plus oral capecitabine 1000 mg/m2 twice a day (BID) (2000 mg/m2 daily dose) x 14 days, followed by 1 week of rest.
- Capecitabine: Capecitabine alone: Capecitabine 1250 mg/m2 BID (2500 mg/m2 daily dose) x 14 days, followed by 1 week of rest.
Period: Overall Study
Arm/Group | Ixabepilone + Capecitabine | Capecitabine
Started | 609 | 612
Completed | 15 (Participants who received 18 or more cycles of treatment.) | 15 (Participants who received 18 or more cycles of treatment.)
Not Completed | 594 | 597
Not completed — Adverse Event | 12 | 17
Not completed — Death | 8 | 18
Not completed — Disease Progression/Relapse | 270 | 388
Not completed — Physician Decision | 50 | 61
Not completed — Lost to Follow-up | 1 | 2
Not completed — Study Drug Toxicity | 179 | 66
Not completed — Withdrawal by Subject | 55 | 30
Not completed — Still On Treatment | 2 | 1
Not completed — Not Treated | 12 | 11
Not completed — Ineligible | 2 | 1
Not completed — Noncompliance | 2 | 1
Not completed — New primary cancer | 1 | 0
Not completed — Impending surgery | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ixabepilone + Capecitabine | Capecitabine | Total
Number analyzed (Participants) | 609 | 612 | 1221
Age, Customized [Number; unit: participants]
  <65 years | 532 | 531 | 1063
  ≥65 years | 77 | 81 | 158
  <50 years | 225 | 235 | 460
  ≥50 years | 384 | 377 | 761
Age, Continuous [Median (Full Range); unit: years] | 53.0 [23.0 to 78.0] | 53.0 [24.0 to 81.0] | 53.0 [23.0 to 81.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 609 | 612 | 1221
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 90 | 69 | 159
  Black or African American | 25 | 21 | 46
  White | 480 | 502 | 982
  Unknown or Not Reported | 13 | 18 | 31
Karnofsky performance Status [Number; unit: units on a scale] — Karnofsky Performance Scale Index measures a patient's functional impairment: 100-80=able to carry on normal activity and work, no special care; 70-50=unable to work; able to live at home and care for most personal needs with assistance; 40=unable to care for self; requires institutional or hospital care. Score reported in multiples of 10.
  units on a scale
    100 | 219 | 265 | 484
    90 | 187 | 188 | 375
    80 | 151 | 130 | 281
    70 | 44 | 26 | 70
    <70 | 2 | 2 | 4
    not reported | 6 | 1 | 7
Menopausal Status [Number; unit: participants]
  Premenopausal | 93 | 90 | 183
  Perimenopausal | 32 | 32 | 64
  Postmenopausal | 475 | 481 | 956
  Not Reported | 9 | 9 | 18
Organ Sites [Number; unit: participants]
  Ascites | 13 | 16 | 29
  Bone | 283 | 287 | 570
  Brain | 0 | 1 | 1
  Breast | 41 | 54 | 95
  Chest Wall Mass | 47 | 38 | 85
  CNS | 1 | 0 | 1
  Cutaneous | 64 | 57 | 121
  Effusion | 7 | 7 | 14
  Intestine | 1 | 1 | 2
  Lymph Node | 236 | 233 | 469
  Mediastinum | 54 | 52 | 106
  Other | 17 | 30 | 47
  Pleura | 86 | 84 | 170
  Subcutaneous | 23 | 24 | 47
  Visceral, Liver | 273 | 276 | 549
  Visceral, Lung | 221 | 217 | 438
  Visceral, Other | 24 | 26 | 50
Presence with at least 1 lesion [Number; unit: participants] | 606 | 612 | 1218

OUTCOME MEASURES:

1. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined for each patient as the time in months from randomization to the date of progression. Patients who died without a reported prior progression were considered to have progressed on their date of death. Patients who did not progress or die were censored on the date of their last tumor assessment.
Time Frame: every 6 weeks (± 3 days) from randomization while on treatment until documented progression
Population: All randomized patients with measurable disease as stratified at the time of randomization; n=480 and n=480 for the 2 treatment groups, respectively. Analysis was conducted once 903 progressions or deaths were observed in 960 participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone + Capecitabine | Capecitabine
Number analyzed (Participants) | 480 | 480
months | 6.24 [5.59 to 6.77] | 4.40 [4.14 to 5.42]
Statistical Analysis 1: Comparison: Ixabepilone + Capecitabine vs Capecitabine; The analysis was conducted when 903 progressions or deaths (446 in combination:457 in capecitabine) were observed in 960 participants; Test type: Superiority or Other; p = .0005, Log Rank; Hazard Ratio (HR) = .79, 95% CI [.69 to .90]

2. Secondary Outcome: Response Rate (RR)
Description: RR=number of patients in that group whose best response is "partial"(30% decrease in the sum of the longest diameter of target lesions) or "complete" (disappearance of all target lesions), according to the 4-item Response Evaluation Criteria in Solid Tumors (RECIST), divided by the total number of response-evaluable participants
Time Frame: every 6 weeks (± 3 days) from randomization while on treatment until documented progression
Population: Response-evaluable participants (all treated participants with the correct diagnosis of adenocarcinoma originating in the breast who had measurable disease as determined at baseline).
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixabepilone + Capecitabine | Capecitabine
Number analyzed (Participants) | 462 | 462
percentage of participants | 43.3 [38.7 to 47.9] | 28.8 [24.7 to 33.2]
Statistical Analysis 1: Comparison: Ixabepilone + Capecitabine vs Capecitabine; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.89, 95% CI [1.44 to 2.50]

3. Secondary Outcome: Duration of Response
Description: Measured from the time RECIST criteria (described in previous outcome measure) were first met for "complete" or "partial" response until first date of documented disease progression or death. Patients who neither relapsed nor died were censored on the date of last tumor assessment. Median w/ 95% CI estimated using Kaplan Meier Product Limit Method.
Time Frame: every 6 weeks (± 3 days) from randomization while on treatment until documented progression
Population: Response-evaluable participants (all treated patients with the correct diagnosis of adenocarcinoma originating in the breast who had measurable disease as determined at baseline)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ixabepilone + Capecitabine | Capecitabine
Number analyzed (Participants) | 200 | 133
Months | 6.1 [5.5 to 7.0] | 6.3 [5.3 to 7.6]

4. Secondary Outcome: Time to Response
Description: Time to response was defined as the time from the first dose of study therapy until measurement criteria were first met for "partial" or "complete" (whichever status was recorded first) per RECIST criteria (a 4-item scale described in the previous outcome measure).
Time Frame: every 6 weeks (± 3 days) from randomization while on treatment until documented progression
Population: as for outcome 3
Measure: Median (Full Range); unit: weeks
Arm/Group | Ixabepilone + Capecitabine | Capecitabine
Number analyzed (Participants) | 200 | 133
weeks | 6.6 [4.7 to 47.9] | 6.6 [4.6 to 59.4]

5. Secondary Outcome: Treatment-Related Safety Summary
Description: Laboratory values, adverse events, and other symptoms were graded using the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTC) Version 3.0
Time Frame: safety was assessed on a continual basis every cycle while on-treatment and every 4 weeks post treatment until toxicities resolved or were deemed irreversible.
Population: All patients who received at least 1 dose of ixabepilone and/or capecitabine. Participants with baseline hepatic impairment (combination arm, n = 50; capecitabine arm, n = 37), defined as Grade ≥2 AST, ALT or Grade ≥1 total bilirubin, were contraindicated due to disproportionate number of toxic deaths observed in study CA163-046.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone + Capecitabine | Capecitabine
Number analyzed (Participants) | 595 | 603
Participants
  Deaths within 30 days of last dose | 19 | 42
  Treatment-related serious adverse events | 125 | 64
  Treatment-related Grade 3-4 adverse events | 458 | 240
  Treatment-related AEs leading to discontinuation | 286 | 66

6. Secondary Outcome: Symptom Assessment Score Changes From Baseline for Functional Assessment of Cancer Therapy-Breast Symptom Index (FBSI)
Description: Quality of life, as measured by the FBSI, an 8-item, participant-reported instrument to measure symptoms. Each item has 5 possible responses ranging from 0 (not at all) to 4 (very much). The scoring was conducted according to the Functional Assessment of Chronic Illness Therapy manual, Version 4; higher scores reflect fewer symptoms.
Time Frame: Baseline and prior to each 21-day cycle of treatment, and at first posttreatment follow-up assessment
Population: Analysis was conducted on all randomized participants on an intent to treat basis. (Note: while table only reports data up to 24 wks, which represents most results, statistical analysis includes ALL assessments through study and follow-up; a few participants were assessed after more than 100 weeks.)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ixabepilone + Capecitabine | Capecitabine
Number analyzed (Participants) | 609 | 612
units on a scale
  Week 3 (n=440; n=429) | -0.5 (13.7) [-0.96 to 0.20] | 0.0 (4.7) [-0.44 to 0.45]
  Week 6 (n=379; n=353) | -0.9 (15.4) [-1.45 to -0.31] | 0.5 (5.0) [0.02 to 1.06]
  Week 9 (n=330; n=283) | -1.5 (17.4) [-2.15 to -0.79] | 0.7 (5.0) [0.06 to 1.24]
  Week 12 (n=283; n=250) | -1.4 (17.3) [-2.06 to -0.64] | 1.1 (5.2) [0.48 to 1.78]
  Week 15 (n=255; n=240) | -1.9 (17.0) [-2.73 to -1.15] | 1.5 (5.0) [0.90 to 2.18]
  Week 18 (n=205; n=202) | -1.3 (15.7) [-2.07 to -0.50] | 1.2 (5.4) [0.41 to 1.89]
  Week 21 (n=166; n=185) | -1.4 (16.8) [-2.36 to -0.37] | 1.7 (5.1) [0.97 to 2.45]
  Week 24 (n=149; n=141) | -1.4 (17.3) [-2.46 to -0.41] | 1.1 (5.4) [0.19 to 1.96]
Statistical Analysis 1: Comparison: Ixabepilone + Capecitabine vs Capecitabine; There was a statistically significant difference between groups in change from baseline FBSI score favoring capecitabine. A mean change from baseline of 2.5 was considered a clinically meaningful difference (minimally important difference or MID). On-treatment mean changes in the FBSI did not reach the MID in either group; Test type: Superiority or Other; p < 0.0001, Wei-Lachin

7. Primary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time in months from randomization until the date of death. For those patients who had not died, survival duration was censored at the last date the patient was known to be alive. Median OS with 95% CI estimated using the Kaplan-Meier Product Limit Method.
Time Frame: from date of randomization until death
Population: Analysis was conducted on all randomized patients on an intent to treat basis. This study required at least 846 events (deaths) to ensure the 2-sided, α = 0.05 level, log-rank test to have 90% power to show a statistically significant difference in OS between treatment groups when the hazard ratio (HR) is 0.8.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone + Capecitabine | Capecitabine
Number analyzed (Participants) | 609 | 612
months | 16.39 [14.95 to 17.91] | 15.64 [13.86 to 17.02]
Statistical Analysis 1: Comparison: Ixabepilone + Capecitabine vs Capecitabine; This primary analysis was a comparison between the 2 treatment arms using a 2-sided, α=0.05 level log-rank test (to reject the null hypothesis of equality of survival). The analysis was conducted when 880 deaths (430 in combination:450 in capecitabine) were observed from the 1221 randomized participants; Test type: Superiority or Other; p = .1162, Log Rank — The test was stratified by (taxane resistance [yes/no], measurable disease versus non-measurable disease, prior chemotherapy for metastatic disease [yes/no], and anthracycline resistance [yes/no]); The analysis was conducted at the 0.05 level and no adjustments were performed; Hazard Ratio (HR) = .90, 95% CI [.78 to 1.03]
Statistical Analysis 2: Comparison: Ixabepilone + Capecitabine vs Capecitabine; This prespecified secondary analysis was a Cox model adjusted for age, Karnofsky performance status, number of organ sites, estrogen receptor status, hepatic impairment, time from diagnosis, liver/lung metastases; Test type: Superiority or Other; p = .0231, Regression, Cox; Hazard Ratio (HR) = .85, 95% CI [.75 to .98]

ADVERSE EVENTS:
Arm/Group | Capecitabine | Ixabepilone + Capecitabine
Serious Adverse Events (participants affected / at risk) | 192/603 | 205/595
Other Adverse Events (participants affected / at risk) | 564/603 | 590/595
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine (N=603) | Ixabepilone + Capecitabine (N=595)
EYE PAIN (Eye disorders) | 1 | 0
ECTROPION (Eye disorders) | 0 | 1
EYELID PTOSIS (Eye disorders) | 1 | 0
VISUAL DISTURBANCE (Eye disorders) | 0 | 1
BLINDNESS UNILATERAL (Eye disorders) | 0 | 1
ULCERATIVE KERATITIS (Eye disorders) | 1 | 0
DIAGNOSTIC PROCEDURE (Investigations) | 1 | 0
HAEMOGLOBIN DECREASED (Investigations) | 0 | 1
BLOOD ALBUMIN DECREASED (Investigations) | 0 | 1
PLATELET COUNT DECREASED (Investigations) | 2 | 2
BLOOD PHOSPHORUS INCREASED (Investigations) | 0 | 1
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 3
PROTHROMBIN TIME PROLONGED (Investigations) | 1 | 0
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 3
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 1
PERICARDITIS (Cardiac disorders) | 1 | 0
ANGINA UNSTABLE (Cardiac disorders) | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | 0 | 1
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 2
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 4 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 | 0
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 | 1
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 0
SHOCK (Vascular disorders) | 1 | 0
PHLEBITIS (Vascular disorders) | 0 | 1
THROMBOSIS (Vascular disorders) | 2 | 2
HYPOTENSION (Vascular disorders) | 1 | 4
LYMPHOEDEMA (Vascular disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 1
THROMBOPHLEBITIS (Vascular disorders) | 1 | 0
VENOUS THROMBOSIS (Vascular disorders) | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 6 | 3
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1 | 0
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 1 | 0
DEPRESSED MOOD (Psychiatric disorders) | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 4 | 2
CHOLANGITIS (Hepatobiliary disorders) | 1 | 0
HEPATIC PAIN (Hepatobiliary disorders) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0
HEPATIC FAILURE (Hepatobiliary disorders) | 3 | 2
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 2 | 0
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 0 | 1
HYPERSENSITIVITY (Immune system disorders) | 0 | 4
ATAXIA (Nervous system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 1 | 1
DYSTONIA (Nervous system disorders) | 0 | 1
EPILEPSY (Nervous system disorders) | 0 | 1
HEADACHE (Nervous system disorders) | 3 | 2
DIZZINESS (Nervous system disorders) | 6 | 0
NEURALGIA (Nervous system disorders) | 0 | 1
CONVULSION (Nervous system disorders) | 0 | 2
MONOPLEGIA (Nervous system disorders) | 1 | 0
SOMNOLENCE (Nervous system disorders) | 1 | 0
HEMIPARESIS (Nervous system disorders) | 1 | 1
PARAESTHESIA (Nervous system disorders) | 0 | 1
HYPOAESTHESIA (Nervous system disorders) | 0 | 1
ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
POLYNEUROPATHY (Nervous system disorders) | 0 | 1
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 | 1
AUTONOMIC NEUROPATHY (Nervous system disorders) | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 | 3
DEMYELINATING POLYNEUROPATHY (Nervous system disorders) | 0 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 6
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1
ILEUS (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 7 | 12
ASCITES (Gastrointestinal disorders) | 1 | 0
COLITIS (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 17 | 24
DIARRHOEA (Gastrointestinal disorders) | 33 | 23
GASTRITIS (Gastrointestinal disorders) | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 2 | 5
CONSTIPATION (Gastrointestinal disorders) | 2 | 6
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1
OESOPHAGITIS (Gastrointestinal disorders) | 0 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 7
PANCREATIC CYST (Gastrointestinal disorders) | 1 | 0
MOUTH ULCERATION (Gastrointestinal disorders) | 1 | 0
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 1
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 1
SEPSIS (Infections and infestations) | 3 | 6
EMPYEMA (Infections and infestations) | 1 | 0
CYSTITIS (Infections and infestations) | 1 | 1
INFECTION (Infections and infestations) | 4 | 4
PNEUMONIA (Infections and infestations) | 5 | 6
CELLULITIS (Infections and infestations) | 1 | 3
ERYSIPELAS (Infections and infestations) | 1 | 0
MENINGITIS (Infections and infestations) | 0 | 1
PARONYCHIA (Infections and infestations) | 0 | 1
ABSCESS LIMB (Infections and infestations) | 1 | 0
LYMPHANGITIS (Infections and infestations) | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 1 | 2
TUBERCULOSIS (Infections and infestations) | 1 | 1
FUNGAL SEPSIS (Infections and infestations) | 1 | 0
NAIL INFECTION (Infections and infestations) | 0 | 1
GASTROENTERITIS (Infections and infestations) | 2 | 1
LOBAR PNEUMONIA (Infections and infestations) | 0 | 1
WOUND INFECTION (Infections and infestations) | 3 | 1
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 0
NEUTROPENIC SEPSIS (Infections and infestations) | 0 | 1
VAGINAL CELLULITIS (Infections and infestations) | 1 | 0
ABDOMINAL INFECTION (Infections and infestations) | 1 | 0
ANORECTAL INFECTION (Infections and infestations) | 0 | 1
BACTERIAL INFECTION (Infections and infestations) | 0 | 1
LOCALISED INFECTION (Infections and infestations) | 0 | 1
NEUTROPENIC INFECTION (Infections and infestations) | 0 | 1
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
CATHETER RELATED INFECTION (Infections and infestations) | 3 | 4
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
GASTROENTERITIS NORWALK VIRUS (Infections and infestations) | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
DYSURIA (Renal and urinary disorders) | 0 | 1
OLIGURIA (Renal and urinary disorders) | 0 | 1
RENAL ATROPHY (Renal and urinary disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 3 | 0
HYDRONEPHROSIS (Renal and urinary disorders) | 1 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 0
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 0 | 1
CATHETER PLACEMENT (Surgical and medical procedures) | 1 | 0
CENTRAL VENOUS CATHETERISATION (Surgical and medical procedures) | 0 | 3
ANOREXIA (Metabolism and nutrition disorders) | 5 | 2
DEHYDRATION (Metabolism and nutrition disorders) | 7 | 7
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 5 | 7
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 8
NEUTROPENIA (Blood and lymphatic system disorders) | 8 | 18
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 | 4
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 5 | 34
RASH (Skin and subcutaneous tissue disorders) | 1 | 3
BLISTER (Skin and subcutaneous tissue disorders) | 0 | 1
PURPURA (Skin and subcutaneous tissue disorders) | 1 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 1
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 1
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN REACTION (Skin and subcutaneous tissue disorders) | 0 | 1
SWELLING FACE (Skin and subcutaneous tissue disorders) | 1 | 0
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 0 | 2
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 | 1
DERMATITIS EXFOLIATIVE (Skin and subcutaneous tissue disorders) | 0 | 1
STEVENS-JOHNSON SYNDROME (Skin and subcutaneous tissue disorders) | 1 | 0
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 3 | 5
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 1
FRACTURE (Injury, poisoning and procedural complications) | 1 | 4
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 7
DRUG TOXICITY (Injury, poisoning and procedural complications) | 1 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 3
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 | 0
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
PUBIC RAMI FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
TRACHEAL OBSTRUCTION (Injury, poisoning and procedural complications) | 0 | 1
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 0 | 1
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 4 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 3
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 2
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 2 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 0 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 25 | 10
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ALVEOLITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 3
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 2
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 13 | 7
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 | 5
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PAIN (General disorders) | 2 | 3
FATIGUE (General disorders) | 6 | 8
PYREXIA (General disorders) | 8 | 6
ASTHENIA (General disorders) | 2 | 1
CHEST PAIN (General disorders) | 2 | 1
HYPOTHERMIA (General disorders) | 0 | 1
SUDDEN DEATH (General disorders) | 1 | 1
EXTRAVASATION (General disorders) | 0 | 1
CATHETER THROMBOSIS (General disorders) | 1 | 0
MULTI-ORGAN FAILURE (General disorders) | 0 | 1
CATHETER SITE OEDEMA (General disorders) | 0 | 1
MUCOSAL INFLAMMATION (General disorders) | 4 | 6
INJECTION SITE EXTRAVASATION (General disorders) | 0 | 1
PERFORMANCE STATUS DECREASED (General disorders) | 1 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 4 | 5
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MALIGNANT ASCITES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BREAST CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 5
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 43 | 17
PERICARDIAL EFFUSION MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine (N=603) | Ixabepilone + Capecitabine (N=595)
WEIGHT DECREASED (Investigations) | 104 | 194
WEIGHT INCREASED (Investigations) | 47 | 26
HAEMOGLOBIN DECREASED (Investigations) | 22 | 44
PLATELET COUNT DECREASED (Investigations) | 13 | 33
NEUTROPHIL COUNT DECREASED (Investigations) | 21 | 67
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 13 | 44
INSOMNIA (Psychiatric disorders) | 37 | 84
HEADACHE (Nervous system disorders) | 73 | 97
DIZZINESS (Nervous system disorders) | 50 | 69
DYSGEUSIA (Nervous system disorders) | 14 | 67
HYPOREFLEXIA (Nervous system disorders) | 17 | 37
PARAESTHESIA (Nervous system disorders) | 45 | 115
NEUROPATHY PERIPHERAL (Nervous system disorders) | 12 | 46
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 23 | 56
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 64 | 258
NAUSEA (Gastrointestinal disorders) | 243 | 315
VOMITING (Gastrointestinal disorders) | 168 | 250
DIARRHOEA (Gastrointestinal disorders) | 244 | 266
DYSPEPSIA (Gastrointestinal disorders) | 45 | 51
STOMATITIS (Gastrointestinal disorders) | 68 | 118
CONSTIPATION (Gastrointestinal disorders) | 73 | 161
ABDOMINAL PAIN (Gastrointestinal disorders) | 77 | 88
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 47 | 55
ANOREXIA (Metabolism and nutrition disorders) | 99 | 183
ANAEMIA (Blood and lymphatic system disorders) | 44 | 69
LEUKOPENIA (Blood and lymphatic system disorders) | 28 | 85
NEUTROPENIA (Blood and lymphatic system disorders) | 49 | 159
RASH (Skin and subcutaneous tissue disorders) | 25 | 68
ALOPECIA (Skin and subcutaneous tissue disorders) | 20 | 245
DRY SKIN (Skin and subcutaneous tissue disorders) | 39 | 51
ERYTHEMA (Skin and subcutaneous tissue disorders) | 12 | 34
PRURITUS (Skin and subcutaneous tissue disorders) | 17 | 31
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 77 | 193
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 75 | 79
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 412 | 383
MYALGIA (Musculoskeletal and connective tissue disorders) | 22 | 146
BACK PAIN (Musculoskeletal and connective tissue disorders) | 62 | 70
BONE PAIN (Musculoskeletal and connective tissue disorders) | 45 | 55
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 30 | 119
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 5 | 30
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 56 | 112
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 37 | 85
COUGH (Respiratory, thoracic and mediastinal disorders) | 68 | 89
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 84 | 99
PAIN (General disorders) | 20 | 32
FATIGUE (General disorders) | 166 | 272
PYREXIA (General disorders) | 66 | 84
ASTHENIA (General disorders) | 72 | 128
OEDEMA PERIPHERAL (General disorders) | 43 | 63
MUCOSAL INFLAMMATION (General disorders) | 53 | 79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.